CLINICAL TRIAL: NCT05089383
Title: Vaginal Versus Combined Use of Progesterone in Fresh IVF/ICSI Cycles
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Collaborators: Iaso Maternity Hospital, Athens, Greece (Other)
Responsible Party: Principal Investigator, Nikos Vlahos, Professor of Obstetrics, Gynecology and Assisted Reproduction, University of Athens
Other Study IDs: ARETAIEION UNIVERSITY HOSPITAL
Record Dates: First submitted 2021-10-10; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Luteal Phase
Keywords: IVF; PROGESTERONE
MeSH Terms: interventions — Utrogestan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- combined progesterone group: patients will receive vaginal plus subcutaneous or per os progesterone
  Interventions: Drug: Utrogestan
- Vaginal progesterone group: patients will receive vaginal progesterone
  Interventions: Drug: Utrogestan

INTERVENTIONS:
Drug: Utrogestan — PROSPECTIVE STUDY
  Other Names: PROLUTEX,VASCLOR

SUMMARY:
Hypothesis: the combined use of progesterone administration for luteal phase support is superior to the single route of progesterone administration in terms of pregnancy outcome parameters in women undergoing fresh IVF/ICSI cycles.

DETAILED DESCRIPTION:
In ART (IVF/ICSI), most of the studies have shown a deficiency of progesterone during the luteal phase, especially due to the use of GnRH analogs. The lack of progesterone leads to abnormal endometrial development and consequently to desynchronization between the latter and the blastocyst implantation. Therefore, it is a standard of care to use progesterone for luteal phase support after embryo transfer and during the first trimester, in case of pregnancy.

According to ESHRE guidelines, either of vaginal, oral, subcutaneous or intramuscular route is advisable.

But, until now, there is no robust evidence on the effect on pregnancy outcome of the combined route of progesterone administration compared to the standard of care (single route).

The aim of this study is to compare the effectiveness of the combined route of progesterone administration to the single route.

The study is a prospective cohort study. Participants will receive either standard treatment with single route (vaginal) progesterone administration according to the ESHRE guidelines, or combination of more than one routes of administration, that is vaginal plus oral or subcutaneous progesterone, starting afterthe fresh embryo transfer until 12 weeks of gestation or a negative pregnancy test.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a documented history of infertility, aged 22-40, undergoing fresh embryo transfer after IVF/ICSI, under informed consent.
* Physiological menstrual cycles (24-35 days), normal endocrine function (FSH ≤ 15 IU / ml), transvaginal ultrasound without pathological findings, free personal medical history, indication for IVF/ICSI.

Exclusion Criteria:

* Endocrine or metabolic disorders, e.g., PCO (S), pathology of the uterus and/or endometrium, basal FSH levels> 15 IU / ml, major surgery in the ovaries (removal), and age <22 years and > 40 years old.
* Active pelvic inflammatory disease
* IVF/ICSI with donor eggs
* Previous participation in this trial

Ages: 22 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Infertile couples with an indication for IVF/ICSI (both Units).
Sampling Method: Probability Sample
Enrollment: 698 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | 9 months]
  The percentage of viable embryo after 20 weeks of gestation
Abortion rate | 20 weeks
  Loss of pregnancy up to 20 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Vlachos, Study Director — National and Kapodistrian University of Athens
Locations (1):
- National and Kapodistrian University of Athens, Athens, Attica, Greece

REFERENCES:
- [Background] van der Linden M, Buckingham K, Farquhar C, Kremer JA, Metwally M. Luteal phase support for assisted reproduction cycles. Cochrane Database Syst Rev. 2015 Jul 7;2015(7):CD009154. doi: 10.1002/14651858.CD009154.pub3. PMID 26148507
- [Background] Practice Committee of the American Society for Reproductive Medicine. Progesterone supplementation during the luteal phase and in early pregnancy in the treatment of infertility: an educational bulletin. Fertil Steril. 2008 Apr;89(4):789-92. doi: 10.1016/j.fertnstert.2008.02.012. PMID 18406835
- [Background] Pabuccu E, Pabuccu R, Gurgan T, Tavmergen E. Luteal phase support in fresh and frozen embryo transfer cycles. J Gynecol Obstet Hum Reprod. 2020 Jun 22:101838. doi: 10.1016/j.jogoh.2020.101838. Online ahead of print. PMID 32585391
- [Background] Tournaye H, Sukhikh GT, Kahler E, Griesinger G. A Phase III randomized controlled trial comparing the efficacy, safety and tolerability of oral dydrogesterone versus micronized vaginal progesterone for luteal support in in vitro fertilization. Hum Reprod. 2017 May 1;32(5):1019-1027. doi: 10.1093/humrep/dex023. PMID 28333318
- [Background] Baker VL, Jones CA, Doody K, Foulk R, Yee B, Adamson GD, Cometti B, DeVane G, Hubert G, Trevisan S, Hoehler F, Jones C, Soules M. A randomized, controlled trial comparing the efficacy and safety of aqueous subcutaneous progesterone with vaginal progesterone for luteal phase support of in vitro fertilization. Hum Reprod. 2014 Oct 10;29(10):2212-20. doi: 10.1093/humrep/deu194. Epub 2014 Aug 6. PMID 25100106
- [Background] Tomic V, Kasum M, Vucic K. The role of luteal support during IVF: a qualitative systematic review. Gynecol Endocrinol. 2019 Oct;35(10):829-834. doi: 10.1080/09513590.2019.1603288. Epub 2019 Apr 29. PMID 31032676
- [Background] Griesinger G, Blockeel C, Sukhikh GT, Patki A, Dhorepatil B, Yang DZ, Chen ZJ, Kahler E, Pexman-Fieth C, Tournaye H. Oral dydrogesterone versus intravaginal micronized progesterone gel for luteal phase support in IVF: a randomized clinical trial. Hum Reprod. 2018 Dec 1;33(12):2212-2221. doi: 10.1093/humrep/dey306. PMID 30304457